CLINICAL TRIAL: NCT03321253
Title: Changes of Macular Pigment Optical Density and Parameters After Nd: YAG Laser Posterior Capsulotomy in Cases With Posterior Capsule Opacification
Brief Title: Changes of Macular Pigment and Parameters of Eyes After YAG Laser Treatment in Cases With Capsule Opacification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyon Kocatepe University Hospital (Other)
Responsible Party: Principal Investigator, Bunyamin Kutluksaman, Principal Investigator, Afyon Kocatepe University Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-2 2017/172
Record Dates: First submitted 2017-10-15; First posted 2017-10-25 (Actual); Results first posted 2019-06-28 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Posterior Capsule Opacification; Retinal Degeneration; Retinal Detachment; Anterior Chamber Angle Congestion; Macula Edema; Macular Pigmentation; Choroid Disease
Keywords: Posterior Capsule Opacification; Macular Pigment Optical Density; Anterior Chamber Parameters; Nd: YAG Laser Posterior Capsulotomy; Posterior Capsulotomy; Cystoid Macular Edema; Choroidal Thickness
MeSH Terms: conditions — Retinal Degeneration; Retinal Detachment; Choroid Diseases; Macular Edema

STUDY DESIGN:
Intervention Model Description: sequential self-controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Nd: YAG laser posterior capsulotomy (Experimental): Posterior capsulotomy was performed by using Nd: YAG laser and macular pigment optical density, intra ocular pressure, choroidal thickness, macular thickness and anterior chamber parameters were measured before Nd: YAG laser, at 1 week, 1 month and 2 months
  Interventions: Device: Nd: YAG laser posterior capsulotomy

INTERVENTIONS:
Device: Nd: YAG laser posterior capsulotomy — Nd: YAG laser posterior capsulotomy
  Other Names: Tango Laserex

SUMMARY:
It has been hypothesized that potential effects of laser Nd: YAG laser posterior capsulotomy may affect macular pigment as well as choroidal thickness, macular thickness and anterior chamber parameters, so it was aimed to investigate possible effects of Nd: YAG laser posterior capsulotomy on macular pigment optical density, choroidal thickness, macular thickness and anterior chamber parameters in cases with posterior capsule opacification in this study.

DETAILED DESCRIPTION:
This clinical trial was conducted following the principles of the Declaration of Helsinki. The local authorized clinical trials ethics committee approved the protocol and consent forms (Afyon Kocatepe University Clinical Trials Ethics Committee, 2011-KAEK-2 2017/172). Between 2015 and 2016, 38 pseudophakic participants were enrolled in this study. After providing information to patients about the disease and treatment, patients predicted to show adherence to treatment, were enrolled in the study.

Detailed ophthalmological examinations of all subjects were performed prior to Nd: YAG laser posterior capsulotomy intervention. Anterior chamber parameters of cases with PCO were measured Measurements of IOP, anterior chamber parameters, visual acuity, Slit-lamp, gonioscopy and fundus examinations, and measurements of central macular thickness (CMT), choroidal thicknesses (CTs), and MPOD were performed after maximal pupil dilatation.

Proposed procedure, including risks, beneﬁts, and alternatives were discussed with all subjects, and all participants signed of informed consent form.

Choroidal thicknesses were recorded as subfoveal CT (SCT), nasal CT (NCT) and temporal CT (TCT).

MPOD measurements were subsequently made by using luminance differential thresholds test. After measurements a refractive surgery specialist carried out Nd: YAG laser posterior capsulotomy interventions to patients who were decided to applying Nd:YAG laser capsulotomy.

All examinations and measurements were repeated and recorded at 1st week, 1st and 2nd month.

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity (BCVA) logMAR <0.3
* Duration at least 2 years after cataract surgery
* Between the ages of 45 and 65 years (45≤age≤65)

Exclusion Criteria:

* Corneal scarring, diffuse posterior PCO or intravitreal hemorrhage that prevents appearance of the fundus
* Occluded angle by gonioscopy (grade 0, narrow angle, grade I, grade II)
* Presence of macular or peripheral retinal pathologies or choroidopathy
* High risk for RD
* Presence of macular edema in the macular area
* Detection of macular fluid or edema in OCT
* Active intraocular inflammation
* Previous laser PRP, Nd: YAG laser posterior capsulotomy, laser iridotomy or selective laser trabeculoplasty interventions
* Previous iridectomy, glaucoma or vitreoretinal surgery
* Glass intraocular lens
* Spherical refractive error ≥ ±6.00 D or cylinder refractive error ≥ ±3.00 D
* Inadequate stability of the eye
* Systemic diseases that may affect the choroidal blood flow such as cardiological diseases
* Current use of carotenoid supplementation
* Changing eating habits
* Gastrointestinal diseases that could cause disturbance of dietary absorption

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-05-16 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.37 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 19
Region of Enrollment [Number; unit: participants]
  Turkey | 38

OUTCOME MEASURES:

1. Primary Outcome: Changes of Foveal and Pericentral Pigment Optical Density (Log Unit) From Baseline at 2 Months
Description: Foveal and pericentral pigment optical density was measured by using color perimetry technique and recorded as log unit before Nd: YAG laser posterior capsulotomy, at 1 week, 1 month and 2 months
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: log unit
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Number analyzed (Participants) | 38
log unit
  MPOD fovea at baseline | 0.55 (0.07)
  MPOD fovea at 1-week | 0.52 (0.08)
  MPOD fovea at 1-month | 0.51 (0.09)
  MPOD fovea at 2-month | 0.5 (0.09)
  MPOD pericentral at baseline | 0.33 (0.05)
  MPOD pericentral at 1-week | 0.31 (0.05)
  MPOD pericentral at 1-month | 0.3 (0.06)
  MPOD pericentral at 2-month | 0.29 (0.06)
Statistical Analysis 1: Comparison: Nd: YAG Laser Posterior Capsulotomy; Test type: Other; p < 0.01, ANOVA

2. Primary Outcome: Changes of Subfoveal, Temporal and Nasal Choroidal Thicknesses (Micrometer) From Baseline at 2 Months
Description: Subfoveal, temporal and nasal choroidal thicknesses were measured by using enhanced-deep imaging optical coherence tomography and recorded as micrometer before Nd: YAG laser posterior capsulotomy, at 1 week, at 1-month and at 2-month
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Number analyzed (Participants) | 38
micrometer
  Subfoveal choroidal thickness baseline | 276.46 (19.36)
  Subfoveal choroidal thickness at 1-week | 276.54 (19.45)
  Subfoveal choroidal thickness at 1-month | 276.86 (19.42)
  Subfoveal choroidal thickness at 2-month | 276.76 (19.36)
  Temporal choroidal thickness at baseline | 275.04 (20.59)
  Temporal choroidal thickness at 1-week | 275.02 (20.67)
  Temporal choroidal thickness at 1-month | 275.23 (20.64)
  Temporal choroidal thickness at 2-month | 275.03 (20.56)
  Nasal choroidal thickness at baseline | 271.16 (19.64)
  Nasal choroidal thickness at 1-week | 271.33 (19.74)
  Nasal choroidal thickness at 1-month | 271.75 (19.71)
  Nasal choroidal thickness at 2-month | 271.74 (19.62)

3. Primary Outcome: Changes of Anterior Chamber Depth (Millimeter) From Baseline at 2 Months
Description: Anterior chamber depth was measured by using anterior segment module optical coherence tomography and recorded as millimeter before Nd: YAG laser posterior capsulotomy, at 1 week, at 1-month and at 2-month
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Number analyzed (Participants) | 38
millimeter
  ACD at baseline | 3.7 (0.06)
  ACD at 1-week | 3.73 (0.06)
  ACD at 1-month | 3.74 (0.06)
  ACD at 2-month | 3.75 (0.07)

4. Primary Outcome: Changes of Iridocorneal Angle From Baseline at 2 Months
Description: Iridocorneal angle was measured by using anterior segment module optical coherence tomography and recorded as millimeter before Nd: YAG laser posterior capsulotomy, at 1 week, at 1-month and 2-month
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Number analyzed (Participants) | 38
degree
  ICA at baseline | 36.59 (1.22)
  ICA at 1-week | 39.92 (2.1)
  ICA at 1-month | 41.62 (3.39)
  ICA at 2-month | 42.04 (4.18)

5. Secondary Outcome: Changes of Central Macular Thicknesses (Micrometer) From Baseline at 2 Months
Time Frame: 2 Months
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
Number analyzed (Participants) | 38
micrometer
  Central Macular Thickness Baseline | 235.79 (13.48)
  Central Macular Thickness 1-week | 243.08 (14.32)
  Central Macular Thickness 1-month | 244.76 (14.82)
  Central Macular Thickness 2-month | 245.5 (15.24)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality, and Serious-Adverse Events were not monitored
Arm/Group | Nd: YAG Laser Posterior Capsulotomy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No